CLINICAL TRIAL: NCT05062590
Title: Socio-geriatric Evaluation (ESOGER): A Clinical Tool in Telehealth to Fight Against Vulnerable Seniors's Health Alterations and Social Isolation
Brief Title: Evolution and Adaptation to Caregiver of a Socio-geriatric Evaluation
Acronym: ESOGER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal (Other Government)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, PhD, Senior researcher, Director of laboratory, Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022-616
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Social Isolation; Aging
MeSH Terms: conditions — Social Isolation | interventions — Health Planning Guidelines

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Intervention (Experimental): Experimental: Group 1 The intervention group will take the ESOGER questionnaire at month 0 and month 3 ( beginning and end) and receive recommendations following their needs.
  Interventions: Other: Recommendations
- Group control (No Intervention): The participants will only take the ESOGER questionnaire at month 0 and month 3 without recommendations

INTERVENTIONS:
Other: Recommendations — Ressources recommendations and interventions curated to the needs of the EP such as refering them to a social activity for socially isolated EP
  Arms: Group Intervention

SUMMARY:
With the COVID-19 pandemic, elderly people (EP) living at home have seen their health deteriorated, thus increasing their needs in support and care. Indeed, while it was estimated that before the pandemic120 000 unattended living at home EP required care and services (taking bath, access to medication and food, etc.), the number doubled after COVID-19. Therefore, the waiting list for socio-medical services for unattended vulnerable clientele without a family doctor grew from 1300 à 1715 EP in a couple of months during the pandemic. With these numbers, it becomes clear that an intervention is needed. Truly, the Institut National d'Excellence en Santé et Services Sociaux (INESSS) conclude that it was pivotal to first identify the most vulnerable EP and second re-orient them according to their needs. Thus the investigator developed the Évaluation et orientation SOcio-GÉRiatrique (ESOGER) questionnaire available on a secure digital plateform enabling both a rapid evaluation and intervention to asses EP needs and provide the adequate ressources. Investigator's previous research has demonstrated that ESOGER is one of the rare clinical tools of first contact in telehealth while being global, multidimensional, and equitable. For this study, the investigator aims to evaluate the effect of ESOGER on EP physical and mental health, loss of autonomy, social isolation, quality of life and ressources consumption.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 and more
* Living at home on the territory CIUSSS-Centre-Sud de l'île-de-Montréal (CCSMTL) of Jeanne-Mance
* Brief Geriatric Assessment (BGA) score of 1/14 or more defining a severly to milidly frail health.

Exclusion Criteria:

* Principal address outside of the CCSMTL's Jeanne-Mance territory
* Participate at another clinical trial, to avoid interferences
* Not understand written or spoken French or English, questionnaires are only available in French and English.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
COVID-19 symptoms | 3 months
  presence or not of fever, cough, and shortness of breath (binary question)
psychological fraility | 3 months
  Anxiety verbal analogic scale, score from 0= no anxiety to 10= extremly anxious
Social health | 3 months
  Issues related to medication and food delivery and access to home care. Presence or not of a shortage in food, medication and home care ( binary question)
Socio-economic characteristics | 3 months
  Presence or not of socio-economic problems (binary questions)
Participant's Quality of life | 3 months
  Measured by the EQ-5D scale with two parts, scale 1 score from 1= no problem to 5 ( sever health problems) and scale 2 visual analogic scale score from 0= worst possible health to 100= best possible health.
Autonomy | 3 months
  ADL scale score from 0= very dependent to 6= very independent and IADL scale score 0= not autonomous 4= autonomous.

SECONDARY OUTCOMES:
Caregiver burden | 3 months
  Based on Zarit scale, score from 0= no burden to 16= high caregiver burnder

CONTACTS AND LOCATIONS:
Locations (1):
- CRIUGM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No